CLINICAL TRIAL: NCT05840887
Title: Knee Osteotomy Associated With Allograft Meniscus Transplantation in Patients With Altered Mechanical Axis, Meniscectomy Outcomes, and Osteoarthritis: Clinical, Biomechanical, and Biological Evaluation
Brief Title: Knee Osteotomy Associated With Allograft Meniscus Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIOMAT
Record Dates: First submitted 2023-04-19; First posted 2023-05-03 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Malalignment, Bone; Osteoarthritis, Knee
Keywords: knee osteotomy; MAT; meniscal allograft transplatation
MeSH Terms: conditions — Bone Malalignment; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: Clinical evaluations will be carried out by medical personnel not involved in treatment to ensure double-blinding
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Ostetomy combined with meniscal allograft transplantation (Experimental): The treatment group will perform osteotomy and meniscal allograft transplantation to restore the meniscal deficiency.
  Interventions: Procedure: Knee osteotomy associated with meniscal allograft transplantation
- Knee Osteotomy (Active Comparator): The control group will consist of patients who will perform an isolated osteotomy.
  Interventions: Procedure: Knee osteotomy

INTERVENTIONS:
Procedure: Knee osteotomy associated with meniscal allograft transplantation — Patients will undergo knee osteotomy associated with meniscal allograft transplantation, which will be implanted by arthroscopic technique with body fixation by all-inside and transosseous sutures to the posterior horn and if necessary to the anterior horn.
  Arms: Knee Ostetomy combined with meniscal allograft transplantation
Procedure: Knee osteotomy — Knee osteotomy
  Arms: Knee Osteotomy

SUMMARY:
This is a prospective randomized double-blind controlled clinical trial with parallel arms and 1:1 allocation.

The main objective of the BIOMAT project is to demonstrate, through an RCT, whether the combined approach by knee osteotomy and MAT can provide clinical improvement over knee osteotomy alone for the treatment of patients with monocompartmental knee OA associated with meniscal insufficiency and lower extremity malalignment. Secondary objectives are to demonstrate whether the addition of MAT to knee osteotomy in patients with monocompartmental OA can improve biomechanical parameters and whether this treatment has protective effects on the joint environment and cartilage degeneration.

DETAILED DESCRIPTION:
Patients with single-compartment arthritic pathology of the knee, axial deviation and meniscal deficit, for whom a surgical indication of corrective osteotomy is placed, will be recruited into the study.

Enrollment takes place during hospitalization and is by the physician. All patients will undergo a knee osteotomy to achieve proper alignment of the lower limb and an arthroscopic procedure to macroscopically verify the status of the cartilage and menisci, with associated minor procedures for surgical cleanup when necessary. After intraoperative confirmation of inclusion criteria (complete meniscal deficit and absence of severe articular cartilage impairment) all patients will undergo synovial biopsy and synovial fluid sampling, half of the patients will also undergo arthroscopic homologous meniscus transplantation.

Clinical, biomechanical and biological evaluations will be performed:

Clinical evaluation of the patient will be done through validated questionnaires before surgery and at 1-3-6-12 months. These will document subjective clinical improvement, functional measurements, and imaging using radiographs as per clinical practice and MRI.

Pitch Analysis will be used for biomechanical assessments, and will be performed before surgery and at 12-month follow-up after surgery for all patients enrolled in the two groups.

basal inflammation will be assessed on synovial tissue and synovial fluid samples collected after intraoperative confirmation of patient inclusion criteria (complete meniscal deficit and absence of severe articular cartilage impairment). Serum/plasma and urine samples will be collected before surgical treatment and at 1-3-6-12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 20 and 60 years;
2. Single-compartment tibiofemoral osteoarthritis (Kellgren-Lawrence grade ≤ 3);
3. Surgical indication of corrective osteotomy (axial deviation of lower extremities > 5°);
4. Meniscal deficit of the compartment affected by the overload due to malalignment;
5. Ability and consent of patients to actively participate in the rehabilitation protocol and clinical and radiological follow-up (RX and MRI)
6. Signature of informed consent

Exclusion Criteria:

1. Patients who are incapacitated or have neurological disorders that may invalidate the research protocol;
2. Diagnosis of neoplastic diseases;
3. Diagnosis of rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis or arthritis resulting from another inflammatory disease; human immunodeficiency virus (HIV) infection, viral hepatitis; chondrocalcinosis;
4. Patients with uncontrolled diabetes mellitus;
5. Patients with uncontrolled thyroid metabolic disorders;
6. Patients abusing alcoholic beverages, drugs or medications;
7. Body Mass Index > 40;
8. Pregnancy or lactation status or intention to become pregnant during the period of study participation;
9. Patients undergoing knee surgery in the previous 12 months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
IKDC-Subjective Score (Subjective International Knee Documentation Committee) | 12 months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function

SECONDARY OUTCOMES:
IKDC-Subjective Score (Subjective International Knee Documentation Committee) | baseline, 1 month, 3 months and 6months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathology. The questionnaire examines 3 categories: symptoms, sports activity, and knee function
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score | baseline, 1 month, 3 months, 6 months and 12 months follow-up
  It's a standardized and widely used questionnaire to assess the condition of patients with knee OA and includes assessment of pain, stiffness and physical function of the joints. It can be administered to the patient. It measures 5 items for pain (range 0-20), two for stiffness (range 0-8), and 17 for functional limitation (range 0-68) that mainly relate to activities of daily living (e.g., getting up from a sitting position, bending over, going up and down stairs etc.); the score is then normalized on a 0-100 scale. Higher values indicated a worse outcome.
KOOS Score ( Knee Injury and Osteoarthritis Outcome score) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  The full questionnaire consists of five subscales and they cover: pain (9 items), symptoms (7 items of which two relate to stiffness), functions and activities of daily living (17 items) physical function, sports activities and leisure (5 items) and quality of life in relation to the knee (4 items). All items in the relevant subscales have the same response mode, use a 5-point Likert scale, and each question is assigned a score from 0 to 4, where 0 indicates "no difficulty" and 4 "a severe difficulty). Score range 0-100 for each subscale
VAS-dolore (Visual Analogue Scale) | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable."
EQ-VAS | baseline, 1 month, 3 months, 6 and 12 months follow-up
  Visual analog scale consisting of a straight line segment (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable."
Tegner Activity Level Scale | baseline, 1 month, 3 months, 6 and 12 months follow-up
  It is a questionnaire to find out the patient's level of physical activity.
Final treatment opinion | 6 and 12 months follow-up
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
WORMS (Whole-Organ Magnetic Resonance Imaging Score) | baseline, 12 months follow-up
  It's a semiquantitative, multifunctional scoring method for knee assessment applicable to conventional MRI techniques.
Kellgren-Lawrence score | baseline, 1 month, 6 months, 12 months follow-up.
  The Kellgren Lawrence scale classifies knee OA into 4 grades of subsequent greater severity, the parameters used being reduced joint space and the presence of osteophytes
Biomechanical analysis | baseline, 12 months follow-up
  Collection of three-dimensional spatial motion data using a 9-camera stereophotogrammetric system combined with wireless 16-channel electromyograph and two force platforms for monitoring foot-ground reaction force. The acquired data will be used to estimate joint rotations and moments, spatiotemporal data, electromyography, and dynamometric data.
Biological assessments | Baseline (pre-operative), 24 hours, 1 month, 3 months, 6 months, 12 months
  Synovial tissue and fluid samples will be collected after intraoperative confirmation of patient inclusion criteria (complete meniscal deficit and absence of severe articular cartilage impairment). Synovial tissue will be fixed, included and analyzed by immunohistochemistry methods for synovitis analysis using a standardized synovitis analysis score (IMSYC). Synovial fluid will be divided into aliquots and stored at -80°C. Inflammatory factors will be analyzed by enzyme immunoassays. Serum/plasma and urine samples will be collected from all patients included in the study at the indicated time points.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
We will be able to share a subset of aggregated data, wich will not allow for the identification of participants.

REFERENCES:
- [Background] Nicolini AP, Christiano ES, Abdalla RJ, Cohen M, de Carvalho RT. Return to Sports After High Tibial Osteotomy Using the Opening Wedge Technique. Rev Bras Ortop (Sao Paulo). 2021 Jun;56(3):313-319. doi: 10.1055/s-0040-1715514. Epub 2020 Sep 25. PMID 34239195
- [Background] McClure PK, Herzenberg JE. The Natural History of Lower Extremity Malalignment. J Pediatr Orthop. 2019 Jul;39(Issue 6, Supplement 1 Suppl 1):S14-S19. doi: 10.1097/BPO.0000000000001361. PMID 31169641
- [Background] Smoak JB, Matthews JR, Vinod AV, Kluczynski MA, Bisson LJ. An Up-to-Date Review of the Meniscus Literature: A Systematic Summary of Systematic Reviews and Meta-analyses. Orthop J Sports Med. 2020 Sep 9;8(9):2325967120950306. doi: 10.1177/2325967120950306. eCollection 2020 Sep. PMID 32953923
- [Background] Liu JN, Agarwalla A, Gomoll AH. High Tibial Osteotomy and Medial Meniscus Transplant. Clin Sports Med. 2019 Jul;38(3):401-416. doi: 10.1016/j.csm.2019.02.006. PMID 31079771
- [Background] Wang K, Sun H, Zhang K, Li S, Wu G, Zhou J, Sun X. Better outcomes are associated with cementless fixation in primary total knee arthroplasty in young patients: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2020 Jan;99(3):e18750. doi: 10.1097/MD.0000000000018750. PMID 32011458
- [Background] Sheng P, Lehto M, Kataja M, Halonen P, Moilanen T, Pajamaki J. Patient outcome following revision total knee arthroplasty: a meta-analysis. Int Orthop. 2004 Apr;28(2):78-81. doi: 10.1007/s00264-003-0526-x. Epub 2003 Nov 20. PMID 15224164
- [Background] Huizinga MR, Gorter J, Demmer A, Bierma-Zeinstra SMA, Brouwer RW. Progression of medial compartmental osteoarthritis 2-8 years after lateral closing-wedge high tibial osteotomy. Knee Surg Sports Traumatol Arthrosc. 2017 Dec;25(12):3679-3686. doi: 10.1007/s00167-016-4232-9. Epub 2016 Jul 7. PMID 27387307
- [Background] Ekhtiari S, Haldane CE, de Sa D, Simunovic N, Musahl V, Ayeni OR. Return to Work and Sport Following High Tibial Osteotomy: A Systematic Review. J Bone Joint Surg Am. 2016 Sep 21;98(18):1568-77. doi: 10.2106/JBJS.16.00036. PMID 27655985
- [Background] Murray R, Winkler PW, Shaikh HS, Musahl V. High Tibial Osteotomy for Varus Deformity of the Knee. J Am Acad Orthop Surg Glob Res Rev. 2021 Jul 9;5(7):e21.00141. doi: 10.5435/JAAOSGlobal-D-21-00141. PMID 34242204
- [Background] Berruto M, Maione A, Tradati D, Ferrua P, Uboldi FM, Usellini E. Closing-wedge high tibial osteotomy, a reliable procedure for osteoarthritic varus knee. Knee Surg Sports Traumatol Arthrosc. 2020 Dec;28(12):3955-3961. doi: 10.1007/s00167-020-05890-0. Epub 2020 Feb 13. PMID 32055878
- [Background] De Bruycker M, Verdonk PCM, Verdonk RC. Meniscal allograft transplantation: a meta-analysis. SICOT J. 2017;3:33. doi: 10.1051/sicotj/2017016. Epub 2017 Apr 21. PMID 29792399
- [Background] Zaffagnini S, Grassi A, Marcheggiani Muccioli GM, Benzi A, Serra M, Rotini M, Bragonzoni L, Marcacci M. Survivorship and clinical outcomes of 147 consecutive isolated or combined arthroscopic bone plug free meniscal allograft transplantation. Knee Surg Sports Traumatol Arthrosc. 2016 May;24(5):1432-9. doi: 10.1007/s00167-016-4035-z. Epub 2016 Feb 9. PMID 26860105
- [Background] Zaffagnini S, Grassi A, Macchiarola L, Stefanelli F, Coco V, Marcacci M, Andriolo L, Filardo G. Meniscal Allograft Transplantation Is an Effective Treatment in Patients Older Than 50 Years but Yields Inferior Results Compared With Younger Patients: A Case-Control Study. Arthroscopy. 2019 Aug;35(8):2448-2458. doi: 10.1016/j.arthro.2019.03.048. PMID 31395185
- [Background] Zaffagnini S, Di Paolo S, Stefanelli F, Dal Fabbro G, Macchiarola L, Lucidi GA, Grassi A. The biomechanical role of meniscal allograft transplantation and preliminary in-vivo kinematic evaluation. J Exp Orthop. 2019 Jun 25;6(1):27. doi: 10.1186/s40634-019-0196-2. PMID 31240420
- [Background] Marcacci M, Zaffagnini S, Kon E, Marcheggiani Muccioli GM, Di Martino A, Di Matteo B, Bonanzinga T, Iacono F, Filardo G. Unicompartmental osteoarthritis: an integrated biomechanical and biological approach as alternative to metal resurfacing. Knee Surg Sports Traumatol Arthrosc. 2013 Nov;21(11):2509-17. doi: 10.1007/s00167-013-2388-0. Epub 2013 Jan 31. PMID 23370980
- [Derived] Zanasi L, Boffa A, De Marziani L, Lisignoli G, Belvedere C, Miceli M, Zaffagnini S, Filardo G, Di Martino A. Knee osteotomy combined with meniscal allograft transplantation versus knee osteotomy alone in patients with unicompartmental knee osteoarthritis: a prospective double-blind randomised controlled trial protocol. BMJ Open. 2024 Dec 12;14(12):e087552. doi: 10.1136/bmjopen-2024-087552. PMID 39672576